CLINICAL TRIAL: NCT00827138
Title: A Multicenter Phase 1 Clinical and Pharmacokinetic Study of DCC-2036 in Subjects With Leukemias (Ph+CML With T315I Mutation Only)
Brief Title: Study Safety and Preliminary Efficacy of DCC-2036 in Patients With Leukemias (Ph+ CML With T315I Mutation)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 2036-01
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — DCC-2036; rebastinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCC-2036 (Experimental): This is a single arm study
  Interventions: Drug: DCC-2036

INTERVENTIONS:
Drug: DCC-2036 — 150 mg BID tablets, continuous dosing of 28 day cycles
  Other Names: rebastinib

SUMMARY:
Rationale: DCC-2036 is a potent broad spectrum inhibitor of BCR-ABL kinase. Inhibition of BCR-ABL has been validated for effective treatment of chronic myeloid leukemia (CML). The emergence of mutant forms of BCR-ABL which resist inhibition by imatinib, dasatinib, and nilotinib is associated with loss of efficacy in treatment of the disease. DCC-2036 is a potent inhibitor of resistant mutants of BCR-ABL including the T315I mutation, and would therefore be expected to effectively treat patients who fail to respond to other BCR-ABL inhibitors. DCC-2036 also inhibits FLT3-ITD, TIE2, KDR, LYN and TRKA kinases. Purpose: to assess the safety and tolerability in patients after continuous administration of DCC-2036 and to determine recommended doses for the conduct of a Phase 2 efficacy trial.

DETAILED DESCRIPTION:
This study will include patients with one of the following: (1) Philadelphia chromosome-positive (Ph+) Chronic myeloid leukemia (CML); (2) FLT3 (gene) internal tandem duplication positive acute myeloid leukemia [FLT3 (gene) ITD-AML]. The investigational drug DCC-2036 has shown in the laboratory to affect different kinds of proteins in CML or AML cancer cells, which may help to stop these cancer cells from growing. This is a Phase 1 study. This Phase 1 study will test the highest safe dose of the investigational drug, DCC-2036, how often the drug should be given, and how well Ph+ CML and AML patients will tolerate DCC-2036. Patients' study doctor will review their past medical history, surgery(s), known allergies, and past/current medications. In addition, blood tests and bone marrow biopsies will be taken to determine if persons are eligible to participate in this study.

During the first part of this study, patients will receive different amounts of DCC-2036 to determine the highest safe dose. Multiple dose levels of DCC-2036 will be tested and as long as no medically unacceptable side effects are noted, the dose will be increased for the next group of study patients. When the highest dose is reached, a larger number of patients will be enrolled to receive DCC-2036 at the highest (safe) dose level. Additional study patients will be enrolled in a group called an "Expansion Group" and receive the study drug at the highest well tolerated dose. Evaluation of the safety and efficacy (how well the study medication treats leukemia) will be studied in this trial. Disease assessment will be monitored as follows: (1) Blood samples will be collected for disease response and for mutational analysis if disease has gotten worse (progressed); (2) Bone marrow samples may be collected by having an area of the hip or chest bone numbed with an anesthetic and a small amount of bone marrow drawn through a needle; (3) For CML patients only, blood samples will be collected for BCR-ABL transcript levels. Patient safety is of primary importance in this Phase 1 study. Safety assessment will be monitored as follows: (1) Physical examinations will be performed regularly during your doctor's visits; (2) Routine blood tests will be performed on a regular basis to assess potential side effects that may be caused by study medication on different organs like (and not limited to) liver, kidney and bone marrow; (3) Based on reports of potential side effects to the heart that may be caused by study medication, patients will be required to have echocardiograms and blood draws to measure the level of serum N-terminal fragment pro B-type natriuretic peptide (NT-proBNP). An echocardiogram is a noninvasive test that uses sound waves to produce images of your heart. These images will tell the doctor how a patient's heart is beating and pumping. The NT-proBNP is a blood test that will help the patient's doctor evaluate how well the heart works. After initial testing is completed, patients will then be required to have these safety evaluations performed at intervals of 3-cycles (approximately every 3 months) for as long as they are taking the study medication. Patients who experience muscle weakness or peripheral neuropathy will be assessed by blood draws to measure creatine phosphokinase (CPK) levels. Measuring CPK levels may help the patient's doctor determine whether or not the symptoms they are experiencing are the result of muscle damage or due to other causes. The most common eye disorders include blurred vision, dry eyes, and visual impairment. Patients will be required to have complete eye (ophthalmologic) evaluations. After initial ophthalmologic exams, patients will be required to have an exam after the completion of every 3 cycles of study medication (approximately every 3 months) and at the time they stop taking study medication. Blood samples will be collected for pharmacokinetic analysis. Pharmacokinetics is the study of the bodily absorption, distribution, metabolism, and excretion of drugs. Blood samples will also be collected for pharmacodynamic analysis. Pharmacodynamic analysis measures biomarkers that are either proteins or genes (also called DNA) that are associated with a disease that may also be related to how you respond to a treatment or what type of side effects may happen. The investigational drug DCC-2036 has not been approved by the United States Food and Drug Administration (FDA). The FDA allows DCC-2036 to be used in research studies only. DCC-2036 will be given to patients only during this study and not after the study is over.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible:

* Ph+ CML in Chronic Phase with T315I mutation
* 18 years or older
* The subject has an ECOG performance status of ≤ 2.
* Adequate organ function as indicated by the following laboratory assessments performed within 14 days prior to the first dose of study drug Hepatic: Serum bilirubin ≤1.5 times upper limit (X ULN) of normal unless due to leukemic involvement or Gilbert's syndrome; aspartate aminotransferase or alanine aminotransferase ≤ 2.5 X ULN; alkaline phosphatase ≤ 2.5 X ULN Renal: Serum creatinine ≤ 1.5 X ULN or 24 hour creatinine clearance ≥ 50 mL/min
* Female subjects of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin pregnancy test within 14 days prior to the start of study drug
* Sexually active subjects who are fertile must agree to use an effective barrier method of contraception while on therapy and for 30 days following discontinuation of study drug. Non-fertile subjects or those not sexually active are also eligible.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria: Subjects presenting with any of the following will not qualify for entry into the study:

* Subject has received chemotherapy or a TKI ≤ 7 days, investigational agent ≤ 14 days, or radiotherapy ≤ 28 days prior to the start of study drug or has not recovered from the acute toxicities associated with any prior treatments including approved therapies, investigational agents, and prior stem cell or bone marrow transplant. The following exceptions apply: i) Hydroxyurea is permitted at any time prior to study enrollment; ii) Glucocorticoids (natural or synthetic) are allowed up to 48 hours prior to the start of the study drug (with the exception of steroids for pre-medication and topical/nasal steroid use which are allowed at any time)
* The subject has AP or BP-CML
* Received immunosuppressive therapy ≤ 28 days prior to the first dose of study drug
* NY Heart Association class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure
* Myocardial infarction within 3 months of the start of study drug
* Active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant
* Any other severe concurrent disease and/or uncontrolled medical conditions, which in the judgment of the investigator, could predispose subjects to unacceptable safety risks or compromise compliance with the protocol
* Human immunodeficiency virus positive
* If female, the subject is pregnant or lactating
* Allergic or hypersensitive to any component of the investigational drug product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of the drug | Completion of the study

SECONDARY OUTCOMES:
Determine the Pharmacokinetic profile and preliminary evidence of clinical response | Completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center; Hedy P Smith, MD, Principal Investigator — Tufts Medical Center; Moshe Talpaz, MD, Principal Investigator — Univ. of Michigan Comprehensive Cancer Center; Kapil Bhalla, MD, Principal Investigator — University of Kansas; Richard A Larson, MD, Principal Investigator — University of Chicago; H.Jean Khoury, MD, Principal Investigator — Emory University; B. Douglas Smith, MD, Principal Investigator — Sidney Kimmel Cancer Center at Johns Hopkins; Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin; David Snyder, M.D., Principal Investigator — City of Hope Medical Center; Javier Pinilla-Ibarz, MD,PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - The University of Kansas Cancer Center, Kansas City, Kansas
  - Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Cortes J, Talpaz M, Smith HP, Snyder DS, Khoury J, Bhalla KN, Pinilla-Ibarz J, Larson R, Mitchell D, Wise SC, Rutkoski TJ, Smith BD, Flynn DL, Kantarjian HM, Rosen O, Van Etten RA. Phase 1 dose-finding study of rebastinib (DCC-2036) in patients with relapsed chronic myeloid leukemia and acute myeloid leukemia. Haematologica. 2017 Mar;102(3):519-528. doi: 10.3324/haematol.2016.152710. Epub 2016 Dec 7. PMID 27927766
- [Derived] O'Hare T, Zabriskie MS, Eiring AM, Deininger MW. Pushing the limits of targeted therapy in chronic myeloid leukaemia. Nat Rev Cancer. 2012 Jul 24;12(8):513-26. doi: 10.1038/nrc3317. PMID 22825216